CLINICAL TRIAL: NCT00000535
Title: Trial of Nonpharmacologic Interventions in Elderly (TONE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Factorial | Purpose: Treatment
Other Study IDs: 78; R01HL048641 (NIH); R01HL048642 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2002-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet, Reducing; Diet, Sodium-Restricted

INTERVENTIONS:
Behavioral: diet, reducing
Behavioral: diet, sodium-restricted

SUMMARY:
To test the efficacy of weight loss and sodium restriction, alone and combined, in maintaining the normotensive state following withdrawal of antihypertensive medications in an elderly cohort. Conducted in collaboration with the National Institute on Aging.

DETAILED DESCRIPTION:
BACKGROUND:

An estimated 30 to 40 percent of elderly persons are treated with blood pressure medications. The efficacy of blood pressure drug therapy in older patients with diastolic or combined diastolic/systolic hypertension is well proven, but such therapy can adversely affect quality of life and biochemical profile. In 1992 when the study started, there was a compelling rationale to identify what proportion of medicated, well-controlled elderly hypertensives could be maintained long-term or greater than 30 months in the normotensive state following withdrawal of blood pressure medications. There was also a need to determine whether nonpharmacologic therapy could significantly increase the proportion with a successful outcome.

DESIGN NARRATIVE:

Randomized. A total of 585 overweight subjects were assigned in a 2 x 2 factorial design to weight loss, sodium reduction, combined weight loss and sodium reduction, or usual life-style control. The remaining 390 subjects of normal weight were assigned in a 2-armed design to a sodium reduction or an attention control group. The control groups were engaged in a series of non-blood pressure related health encounters designed to control for non-specific effects of groups contacts. Withdrawal of antihypertensive medication was attempted following three months of intervention. The primary endpoint was a blood pressure of 150/90 mm Hg or greater, resumption of antihypertensive drug therapy, or the occurrence of a blood pressure-related clinical complication during two to three years of follow-up. Recruitment ended in June, 1994. Follow-up ended in December, 1995. NHLBI support for the trial ended in March, 1997. The NIA supported the Coordinating Center and two clinical centers through February 1998.

The study completion date listed in this record was obtained from the "Completed Date" entered from the old format in the Protocol Registration and Results System (PRS).

ELIGIBILITY:
Men and women with a systolic blood pressure of less than 145 mm Hg and diastolic blood pressure of less than 85 mm Hg on single-drug therapy.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-04; Study Completion 1997-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ettinger — Bowman Gray School of Medicine
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Bowman Gray School of Medicine, Winston-Salem, North Carolina
  - University of Tennessee, Memphis, Tennessee

REFERENCES:
- [Background] Appel LJ, Espeland M, Whelton PK, Dolecek T, Kumanyika S, Applegate WB, Ettinger WH Jr, Kostis JB, Wilson AC, Lacy C, et al. Trial of Nonpharmacologic Intervention in the Elderly (TONE). Design and rationale of a blood pressure control trial. Ann Epidemiol. 1995 Mar;5(2):119-29. doi: 10.1016/1047-2797(94)00056-y. PMID 7795830
- [Background] Espeland MA, Kumanyika S, Kostis JB, Algire J, Applegate WB, Ettinger W, Whelton PK, Bahnson J. Antihypertensive medication use among recruits for the Trial of Nonpharmacologic Interventions in the Elderly (TONE). J Am Geriatr Soc. 1996 Oct;44(10):1183-9. doi: 10.1111/j.1532-5415.1996.tb01367.x. PMID 8855996
- [Background] Whelton PK, Appel LJ, Espeland MA, Applegate WB, Ettinger WH Jr, Kostis JB, Kumanyika S, Lacy CR, Johnson KC, Folmar S, Cutler JA. Sodium reduction and weight loss in the treatment of hypertension in older persons: a randomized controlled trial of nonpharmacologic interventions in the elderly (TONE). TONE Collaborative Research Group. JAMA. 1998 Mar 18;279(11):839-46. doi: 10.1001/jama.279.11.839. PMID 9515998
- [Background] Whelton PK, Babnson J, Appel LJ, Charleston J, Cosgrove N, Espeland MA, Folmar S, Hoagland D, Krieger S, Lacy C, Lichtermann L, Oates-Williams F, Tayback M, Wilson AC. Recruitment in the Trial of Nonpharmacologic Intervention in the Elderly (TONE). J Am Geriatr Soc. 1997 Feb;45(2):185-93. doi: 10.1111/j.1532-5415.1997.tb04505.x. PMID 9033517
- [Background] Kostis JB, Espeland MA, Appel L, Johnson KC, Pierce J, Wofford JL. Does withdrawal of antihypertensive medication increase the risk of cardiovascular events? Trial of Nonpharmacologic Interventions in the Elderly (TONE) Cooperative Research Group. Am J Cardiol. 1998 Dec 15;82(12):1501-8. doi: 10.1016/s0002-9149(98)00694-8. PMID 9874055
- [Background] Kostis JB, Wilson AC, Shindler DM, Cosgrove NM, Lacy CR. Persistence of normotension after discontinuation of lifestyle intervention in the trial of TONE. Trial of Nonpharmacologic Interventions in the Elderly. Am J Hypertens. 2002 Aug;15(8):732-4. doi: 10.1016/s0895-7061(02)02942-4. PMID 12160197
- [Background] Kostis JB, Wilson AC, Hooper WC, Harrison KW, Philipp CS, Appel LJ, Espeland MA, Folmar S, Johnson KC; TONE Cooperative Research Group. Trial Of Nonpharmacologic interventions in the Elderly. Association of angiotensin-converting enzyme DD genotype with blood pressure sensitivity to weight loss. Am Heart J. 2002 Oct;144(4):625-9. doi: 10.1067/mhj.2002.123570. PMID 12360157
- [Background] Kumanyika SK, Espeland MA, Bahnson JL, Bottom JB, Charleston JB, Folmar S, Wilson AC, Whelton PK; TONE Cooperative Research Group. Ethnic comparison of weight loss in the Trial of Nonpharmacologic Interventions in the Elderly. Obes Res. 2002 Feb;10(2):96-106. doi: 10.1038/oby.2002.16. PMID 11836455
- [Background] Appel LJ, Espeland MA, Easter L, Wilson AC, Folmar S, Lacy CR. Effects of reduced sodium intake on hypertension control in older individuals: results from the Trial of Nonpharmacologic Interventions in the Elderly (TONE). Arch Intern Med. 2001 Mar 12;161(5):685-93. doi: 10.1001/archinte.161.5.685. PMID 11231700
- [Derived] Juraschek SP, Cluett JL, Belanger MJ, Anderson TS, Ishak A, Sahni S, Millar C, Appel LJ, Miller ER, Lipsitz LA, Mukamal KJ. Effects of Antihypertensive Deprescribing Strategies on Blood Pressure, Adverse Events, and Orthostatic Symptoms in Older Adults: Results From TONE. Am J Hypertens. 2022 Apr 2;35(4):337-346. doi: 10.1093/ajh/hpab171. PMID 34718403
- [Derived] Chen L, Zhang Z, Chen W, Whelton PK, Appel LJ. Lower Sodium Intake and Risk of Headaches: Results From the Trial of Nonpharmacologic Interventions in the Elderly. Am J Public Health. 2016 Jul;106(7):1270-5. doi: 10.2105/AJPH.2016.303143. Epub 2016 Apr 14. PMID 27077348
- [Derived] Shea MK, Nicklas BJ, Houston DK, Miller ME, Davis CC, Kitzman DW, Espeland MA, Appel LJ, Kritchevsky SB. The effect of intentional weight loss on all-cause mortality in older adults: results of a randomized controlled weight-loss trial. Am J Clin Nutr. 2011 Sep;94(3):839-46. doi: 10.3945/ajcn.110.006379. Epub 2011 Jul 20. PMID 21775558